CLINICAL TRIAL: NCT06243835
Title: A Phase 1a Randomized, Double-blind, Placebo-controlled, Single Site, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of Kindolor Tosylate in Healthy Adults
Brief Title: A Study to Test the Effects of Kindolor at Different Doses in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by sponsor due to low drug bioavailability; no safety concerns were noted.
Sponsor: Lohocla Research Corporation (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIND-2022-01; UH3DA047680 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Kindolor Cohort 1 (Experimental): Kindolor Tosylate
  1 tablet dose 100mg NPO for 8hrs x1 AM PO ex aq
  Interventions: Drug: Kindolor Tosylate
- Kindolor Cohort 2 (Experimental): Kindolor Tosylate tablet
  1 tablet dose 300mg NPO for 8hrs x1 AM PO ex aq
  Interventions: Drug: Kindolor Tosylate
- Kindolor Cohort 3 (Experimental): Kindolor Tosylate
  3 tablets dose 300mg NPO for 8hrs x1 AM PO ex aq
  Interventions: Drug: Kindolor Tosylate
- Kindolor Cohort 4 (Experimental): Kindolor Tosylate
  6 tablets dose 300mg NPO for 8hrs x1 AM PO ex aq
  Interventions: Drug: Kindolor Tosylate
- Placebo Comparator (Placebo Comparator): Placebo to Match tablet(s) NPO for 8hrs x1 AM PO ex aq
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kindolor Tosylate — Kindolor Tosylate enteric coated tablets containing the specified amount of drug product
  Other Names: DCUKA
  Arms: Kindolor Cohort 1; Kindolor Cohort 2; Kindolor Cohort 3; Kindolor Cohort 4
Drug: Placebo — Placebo enteric coated tablets identically matched to the Kindolor Tosylate tablets with equal amount of Prosolv SMCC replacing the Kindolor Tosylate
  Other Names: Placebo to Match
  Arms: Placebo Comparator

SUMMARY:
The goal of this study is to test Kindolor in healthy adults. The main questions it aims to answer are:

* What is the safe dose of Kindolor in healthy volunteers?
* How is Kindolor metabolized by the human body?

Participants will undergo medical tests before and after receiving Kindolor or a placebo to see if there is any difference between the groups.

DETAILED DESCRIPTION:
Eligible participants will undergo intake procedures and baseline evaluations at the clinic the day before dosing. The next day, participants will be randomized to, and receive, either Kindolor tablets or placebo tablets (4 cohorts of escalating doses of Kindolor with 6 Kindolor participants and 2 placebo participants in each cohort). Participants will remain in the clinic for at least an additional 48-hours for safety assessments and blood collections to determine plasma levels of Kindolor, then will be discharged from the clinic and return for follow-up safety tests 7 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteer, ages 18-to-55 years, inclusive.
2. BMI must be between 18 and 32 kg/m2 (inclusive) and weigh a minimum of 50 kg (110 lbs). BMI is calculated as weight in kg divided by the square of height measured in meters.
3. A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
4. If female, be postmenopausal (at least 2 years prior to dosing), surgically sterile (6 months post tubal ligation), or agree to use an acceptable form of birth control from screening until 28 days after dosing. Subjects who claim postmenopausal status will have status confirmed with a follicle-stimulating hormone (FSH) test. Acceptable forms of birth control for females include the following:

   * Vasectomized partner (at least 6 months prior to dosing)
   * Surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to dosing
   * Non-surgical permanent sterilization (eg, Essure procedure) at least 3 months prior to dosing
   * Double barrier (diaphragm with spermicide; condoms with spermicide)
   * Nonhormonal intrauterine device
   * Abstinence (must agree to use a double barrier method if they become sexually active during the study)
5. If male, agree to use an acceptable method of birth control during the study and in the 90 days following dosing. Acceptable forms of birth control for males include the following:

   * Vasectomy (at least 6 months before dosing)
   * Partner is surgically sterilized (see methods above for females)
   * Partner uses oral, injectable, or implantable hormonal contraceptives or intrauterine device (IUD)
   * Double barrier (partner uses diaphragm with spermicide; condoms with spermicide)
   * Abstinence (subject must agree to use a double barrier method if subject becomes sexually active during the study)
6. If female, agree to not breastfeed or donate ova from the time of consenting to the study and for 28 days after dosing the study drug.
7. If male, agree to not donate sperm from the time of consenting to the study and for 90 days after dosing the study drug.
8. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English.
9. Complete all assessments required at screening and baseline and be available to stay in the Phase I unit for a period of approximately 3 days and 2 nights and return for a follow-up visit.
10. Provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
11. Be someone who in the opinion of the investigator would be expected to complete the study protocol.

Exclusion Criteria:

1. History of significant sensitivity to any drug.
2. Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements (including cannabis and cannabis derived products, including CBD-containing products) on a regular basis or use of any of the above within the 2 weeks or 5 half-lives of the respective medication prior to study drug administration.
3. More than moderate alcohol consumption in the past 8 weeks. Moderate alcohol consumption is defined as limiting intake to 2 drinks or less in a day for men and 1 drink or less per day for women. Examples of one drink include: Beer: 12 fluid ounces (355 milliliters); Wine: 5 fluid ounces (148 milliliters); Distilled spirits (80 proof): 1.5 fluid ounces (44 milliliters).
4. Has a clinically significant laboratory test that is out of range of normal limits. An out of range of normal limit laboratory value is clinically significant if associated with one of the following: a) clinical diagnosis; b) systemic signs and symptoms; c) physical exam finding; d) more than 10% above the upper or below the lower limit of normal.
5. Have a urine toxicology screen positive during screening or baseline for any of the following substances:

   1. ethylglucuronide (alcohol metabolite),
   2. amphetamines,
   3. barbiturates,
   4. benzodiazepines,
   5. buprenorphine,
   6. cocaine,
   7. fentanyl,
   8. methylenedioxymethamphetamine (MDMA),
   9. methadone,
   10. methamphetamines,
   11. morphine,
   12. opioids,
   13. oxycodone,
   14. phencyclidine and/or
   15. tetrahydrocannabinol (THC)
6. If female, positive pregnancy test or nursing.
7. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCV Ab) or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening, and the results will be maintained confidentially by the study site.
8. Positive SARS-CoV-2 antigen test prior to 72 hours of clinic intake.
9. History of any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, endocrine, dermatological, metabolic, neurological (nerve injury) or psychiatric disease or disorder, or any uncontrolled medical illness.
10. History of gastroesophageal reflux disease, gastrointestinal ulcers, gastrointestinal bleeding, inflammatory bowel disease or gastroesophageal surgery.
11. Use of any known strong CYP3A4 inhibitors (e.g., ketoconazole) or dual CYP3A4 and 2C9 inhibitor (eg. Fluconazole), or dual CYP3A4 and 2C9 inducer (eg. Rifampin), or use of any monoamine oxidase inhibitors (MAOIs) within 1 month prior to study drug administration.
12. Receipt of any drug by injection within 30 days prior to study drug administration.
13. History of head trauma with loss of consciousness, history of epilepsy, seizures or convulsions, including febrile, alcohol, or drug withdrawal seizures.
14. A clinically notable vital sign abnormality including a history of syncopal or near syncopal events following abrupt change in posture.
15. Have any of the following at screening or baseline:

    * Blood pressure: systolic >140 mmHg, diastolic >90 mmHg at Screening or Day -1.
    * Heart rate: >100 beats/minute at screening or Day -1
16. History of cardiovascular abnormality, including left ventricular dysfunction, sick sinus syndrome, family history of long-QT syndrome, or unexplained sudden deaths in their family.
17. Has a clinically significant abnormal ECG or an ECG with a QTc interval corrected for heart rate using the Fridericia formula (QTcF) > 430 msec.
18. History of gastric surgery, vagotomy, bowel resection, or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption.
19. Has an estimated creatinine clearance (CrCl) outside of normal range.
20. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
21. Receipt of any investigational product within 6 weeks prior to study drug administration.
22. Consumption of alcohol within the 1-day period prior to study drug administration.
23. Consumption of grapefruit or grapefruit products from 3 days prior to study drug administration to study drug administration.
24. Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
25. Current enrollment in another clinical study.
26. Previous enrollment in this study.
27. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive kindolor tosylate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence, Severity and Relationship of Adverse Events [Safety and Tolerability] | From baseline to Day 7
  Changes in clinical laboratory tests, ECG, fecal occult blood tests, vital signs and urine output

SECONDARY OUTCOMES:
Pharmacokinetic AUCt of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  Area under the plasma concentration-time (AUCt) curve from time 0 to the time (t) of last quantifiable concentration (Ct).
Pharmacokinetic AUC∞ of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  Area under the plasma concentration-time curve (AUC∞) from time 0 extrapolated to infinity.
Pharmacokinetic Cmax of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  The maximum observed plasma concentration.
Pharmacokinetic Tmax of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  The observed time to reach maximum plasma concentration.
Pharmacokinetic λz of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  The terminal-phase exponential rate constant.
Pharmacokinetic t1/2 of Kindolor Tosylate | Pre-dose to 48 hours post-dose
  The apparent terminal exponential half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, MD, Principal Investigator — University of California, San Diego
Locations (1):
- The Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No